CLINICAL TRIAL: NCT07136155
Title: Indirect Pulp Capping Versus Hall Crown Technique for the Management of Deep Dentinal Caries of Primary Molars: A Randomized Controlled Trial.
Brief Title: Indirect Pulp Capping Versus Hall Crown Technique for the Management of Deep Dentinal Caries of Primary Molars.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 414 - 2024; 20240506 (Other Grant/Funding Number: Jordan University of Science and Technology)
Record Dates: First submitted 2025-05-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries
Keywords: Dental caries; Hall technique; Indirect pulp capping; primary molars
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall Crown Technique (Experimental): preformed metal crowns (PMCs) cemented with no local anesthesia, caries removal or tooth preparation in one side.
  Interventions: Procedure: Hall Technique
- Indirect pulp capping (Experimental): Selective caries removal to firm dentin followed by placing RMGI base material and subsequent preformed metal crown (PMC)
  Interventions: Procedure: Indirect pulp capping

INTERVENTIONS:
Procedure: Hall Technique — preformed metal crowns (PMCs) cemented with no local anesthesia, caries removal or tooth preparation in one side.
  Arms: Hall Crown Technique
Procedure: Indirect pulp capping — Selective caries removal to hard dentin followed with G.I base material and subsequent preformed metal crown (PMC).
  Arms: Indirect pulp capping

SUMMARY:
This is a randomized clinical trial that aims to compare the clinical and radiographic success of Hall technique (HT) versus Indirect pulp capping (IPC) for the management of deep dentinal caries in primary molars and to compare the child and parent acceptance of HT versus IPC for the management of deep dentinal caries in primary molars.

DETAILED DESCRIPTION:
This is a randomized clinical trial that aims to compare the clinical and radiographic success of Hall technique (HT) versus Indirect pulp capping (IPC) for the management of deep dentinal caries in primary molars and to compare the child and parent acceptance of HT versus IPC for the management of deep dentinal caries in primary molars.

Children aged 4-9 years old presenting with occlusal or proximal carious lesions of primary molars radiographically extending into the inner third or quarter of dentin will be invited to participate in this study. Patients will be randomized into two treatment groups using online block randomization technique (block of 6) and sealed envelope techniques. Time taken for clinical procedure will be recorded by a research assistant prospectively from the time the child sits on the dental chair till the end of procedure. Child pain perception will be recorded during intervention by a blinded research assistant using the Sound Eye Motor scale (SEM). Parental preference and child acceptance for each procedure will be recorded immediately after treatment using parent and child questionnaires. Clinical and radiographic success, and patient satisfaction will be evaluated at 6 and 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Fit and healthy.
* Occlusal or proximal carious lesions on primary molars radiographically extending into the inner third or quarter of dentin.
* Vital pulp with no signs or symptoms of irreversible pulpitis, necrosis, or an abscess.
* No tenderness to percussion, or pathological mobility.
* No radiographic evidence of interradicular/ periapical radiolucency.
* Radiographic evidence of a radiopaque dentin layer between the radiolucent caries lesion and the dental pulp
* Tooth is restorable.
* Patient has good level of cooperation for the intended procedure.
* Parents consented for their children to be included in the study.

Exclusion Criteria:

* Medically compromised children.
* Irreversible pulpitis or pulp necrosis.
* Soft and/or hard tissue pathology.
* Furcal/ periapical pathology.
* Root resorption exceeding one third of the root.
* Pathological mobility.
* Patient has poor level of cooperation for the intended procedure

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient pain perception | Perioperatively
  will be evaluated by an observer (research assistant who will be trained, calibrated, and blinded to the treatment used) and recorded using the Sound, Eyes, and motor scale (SEM);Based on the intensity of the child's discomfort, each parameter is scored into one of four categories (comfort (score 0), mild discomfort (score 1), moderately painful (score 2), and painful (score 3)). The total score can range from 0 to 9, with 9 indicating the highest level of discomfort.
Rate of Radiographic Success | 6,12 months
  Absence of radiographic pathology in the root and the bone in the inter-radicular area.
Child acceptance of treatment | immediately following intervention
  Self-reported child acceptance using questionnaire
Parent acceptance of treatment | immediately following intervention
  Parental acceptance using questionnaire
Rate of Clinical Success | 3,6,12 months
  Absence of clinical symptoms of spontaneous pain, pain on percussion, pathologic mobility or abscess formation.,assessed through taking pain history and clinical examination.

SECONDARY OUTCOMES:
Time taken for intervention | Perioperative/Periprocedural: from the moment the child sits in the chair until the intervention is completed.
  Time taken for providing the intervention, measured in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided